CLINICAL TRIAL: NCT05649553
Title: The Effect of Diabetes Education Given to Children With Type 1 Diabetes Mellitus With Digital Games and Video Animation on Quality of Life
Brief Title: The Effect of Diabetes Education Digital Games and Video Animation on Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Gamze Tınmaz Pehlivan, PhD, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GPehlivan; Sebahat ALTUNDAĞ, Assoc. Prof. (Other: Pamukkale University)
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes education; digital game; video animation
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This study is a parallel group randomized controlled study
Who Masked: Participant
Masking Description: Single blinding was provided that included inclusion criteria and agreement to participate in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Experimental: Intervention Group Application of the Introductory Information Form and the "Quality of Life Scale in Children with Diabetes Mellitus (PedsQL 3.0 Diabetes Scale)" test Giving digital game and video animation-based diabetes education to the children in the experimental group, in addition to the education given by the diabetes nurse, Applying the first post-training follow-up test to children in the experimental and control groups 3 months after the training.
  Applying the post-training-2nd follow-up test to the children in the experimental and control groups 6 months after the training.
  Interventions: Behavioral: digital game and video animation based diabetes education
- Control Group (No Intervention): The control group received routine nursing care in the endocrine policlinic.

INTERVENTIONS:
Behavioral: digital game and video animation based diabetes education — While creating the digital game and video animation, an agreement was made with a software company and this company was responsible for the software and repair of the game. Digital games and video animations cover the basic educational topics of Type 1 diabetes. Expert opinions were received from experts in the field of Child Health and Disease Nursing to ensure the suitability of the content of the educational material. The name of the game site and how to use it were explained to the children in the intervention group by the researcher. In addition, children in the intervention group were given usernames and passwords to log in to the site. Game Sections; What is Diabetes? Medical Nutrition Treatment in Diabetes, Insulin Treatment and Application, Exercise and Physical Activity in Diabetes, Complications of Type 1 Diabetes Mellitus, Diabetes Management at School.
  Other Names: digital game, video animation
  Arms: Intervention Group

SUMMARY:
This research will be conducted to evaluate the effect of digital game and video animation-based diabetes education on the quality of life of children with Type 1 Diabetes. HbA1c, diabetes knowledge and Quality of Life Scale in Children with Diabetes (PedsQL 3.0) score will be taken into consideration when evaluating the quality of life of children with type 1 diabetes.

DETAILED DESCRIPTION:
This research was conducted to examine the effects of diabetes education given to children with Type 1 Diabetes Mellitus with digital game and video animation on quality of life and metabolic control. The study is a single-blind, randomized controlled trial. It was conducted with a total of 55 children with Type 1 Diabetes Mellitus, including the experimental (n=27) and control group (n=28). Diabetes education was given to the experimental group with digital games and video animations. Data were collected before the training, at the 3rd and 6th months after the training. Research data were collected with "Descriptive Information Form", "Quality of Life Scale in Children with Diabetes Mellitus" and "Metabolic Control Parameters Follow-up Form". Children in the control group received routine outpatient examination/check-up and diabetes education by a diabetes nurse. Children in the intervention group were given digital game and video animation-based training, as well as routine outpatient examination/check-up and training given by a diabetes nurse.

ELIGIBILITY:
Inclusion Criteria:

* Children's willingness to participate in the research (written consent of their parents, verbal consent was obtained from the children),
* Being between the ages of 8-12,
* Having been diagnosed with Type 1 Diabetes Mellitus at least 1 year ago
* To have regular follow-ups,
* No communication disability (speech, hearing, vision problems)
* It means having a device (computer) with internet connection at home and being able to use it.

Exclusion Criteria:

* Having any chronic disease together with diabetes,
* Using an insulin pump

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline, 3. and 6. months
  Measuring the changes in HbA1c levels of children with type 1 diabetes before training and at the 3rd and 6th months after training.

SECONDARY OUTCOMES:
Changes in quality of life | Baseline, 3. and 6. months
  Measuring the changes in quality of life of children with type 1 diabetes before training and at the 3rd and 6th months after training.

CONTACTS AND LOCATIONS:
Overall Officials: Sebahat ALTUNDAĞ, AssocProfDr., Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No